CLINICAL TRIAL: NCT03189212
Title: Feasibility Study of Telemedicine for Dialysis Patients Awaiting Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-02146
Record Dates: First submitted 2017-05-31; First posted 2017-06-16 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: End Stage Renal Disease; Kidney Disease, Chronic
Keywords: Telemedicine
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Visit (Active Comparator)
  Interventions: Behavioral: Usual Care Visit
- Telemedicine Visit (Experimental)
  Interventions: Behavioral: Telemedicine Visit

INTERVENTIONS:
Behavioral: Usual Care Visit — Routine 6-month follow up appointment at the NYULMC transplant center
  Arms: Usual Care Visit
Behavioral: Telemedicine Visit — TM visit conducted at the patient's dialysis unit as a replacement to usual 6 month routine f/u visit
  Arms: Telemedicine Visit

SUMMARY:
The purpose of this study is to determine whether a telemedicine follow-up visit at the NYU Langone Transplant Institute is a feasible and acceptable alternative to a traditional in-center follow-up visit.

DETAILED DESCRIPTION:
A six-month prospective randomized-controlled clinical pilot study to evaluate a new intervention for the transplant program: telemedicine (TM) visits. Researchers will target patients on the transplant waiting list who are currently undergoing dialysis. Currently, there are 234 patients on the transplant waiting list who receiving care at dialysis centers in the New York City area. Researchers will select the 10 dialysis centers having the highest number of patients on the transplant list in order to yield a target sample of 45.

Eligible participants will be randomized to 1 of 2 groups: (1) usual care (UC) which is the routine 6-month follow up appointment at the NYULMC transplant center or (2) TM visit conducted at the patient's dialysis unit as a replacement to usual 6 month routine f/u visit. Patients will be followed for 4 months post randomization to determine the number of days that elapse between randomization and routine transplant evaluation. As new clinic appointments are currently experiencing 80-day wait, a 4-month follow-up should be more than adequate to evaluate this primary outcome.

The intervention will be evaluated primarily in terms of efficiency, and secondarily in terms of patient/physician experiences, changes in waiting list status, and referral for living donation.

ELIGIBILITY:
Inclusion Criteria:

* Receiving thrice-weekly hemodialysis treatment for 6 months
* On NYULMC kidney transplant wait list

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Unable to read or otherwise use an iPad (e.g. blind)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
Waiting time | 4 Months
  The study is powered to evaluate wait time for the next transplant clinic appointment, abstracted from the patient's electronic record at the conclusion of the study.
Missed visits | 4 Months
  Using the medical record, researchers will capture the frequency of no-shows, cancellations, and rescheduled visits. At the 4-month time point, researchers will interview patients to collect qualitative data regarding the reasons for missed or rescheduled appointments. They will also collect data regarding the frequency with which TM visits result in transplant coordinator requests for an additional in-person appointment in order to conduct a physical assessment.
Cost | 4 Months
  Researchers will estimate cost of UC and TM in terms of costs borne by the patient (transportation, childcare, missed employment time, missed leisure) using an investigator-developed instrument. They will estimate health care service delivery costs using standard accounting methods to estimate facility costs, wage and fringe rates for staff involved in care (including receptionist, nurse, TM staff), and technology costs (including the iPads, data plans, maintenance and replacement costs).

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Ali, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States